CLINICAL TRIAL: NCT05995418
Title: Monetary Costs of Alzheimer's Disease in China: Protocol for a Cluster-randomized Observational Study
Brief Title: Study on the Health Economic Burden of Alzheimer's Disease in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2023132
Record Dates: First submitted 2023-07-30; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- amnestic mild cognitive impairment(aMCI）: 1. aMCI diagnostic criteria of National Institute of Aging and National Association of Alzheimer's Disease (NIA-AA).
  2. The ClinicalDementiaRating scale (CDR) is 0.5.
  3. Mini-MentalStateExamination (MMSE): MMSE≥17 for those with 0 years of education, ≥20 for those with less than 7 years, and ≥24 for those with more than 7 years.
  4. Memory impairment is prominent, and it may also be accompanied by functional impairment of other cognitive domains.
  5. The onset is insidious and the progress is slow.
  6. Not up to the level of dementia
  Interventions: Other: There was no intervention as this was an observational study.
- mild to moderate AD: Clinical dementia rating (CDR) was used to assess and determine the degree of cognitive impairment of the patients, according to the CDR score, where the mild AD group with a CDR score of 1, and the moderate to severe AD group with a score of 2 to 3.
  Interventions: Other: There was no intervention as this was an observational study.
- severe AD: Clinical dementia rating (CDR) was used to assess and determine the degree of cognitive impairment of the patients, according to the CDR score, where the mild AD group with a CDR score of 1, and the moderate to severe AD group with a score of 2 to 3.
  Interventions: Other: There was no intervention as this was an observational study.

INTERVENTIONS:
Other: There was no intervention as this was an observational study. — There was no intervention as this was an observational study.

SUMMARY:
This study is a multi-center and cross-sectional study. Using standardized case report forms, we randomly selected suitable patients from the cognitive centers of provincial administrative units in Chinese mainland to conduct a questionnaire survey, so as to obtain relevant information about their economic burden.

DETAILED DESCRIPTION:
Under the policy background of building a national cognitive center, this study collected and evaluated the socio-demographic characteristics, geographical location, regional socio-economic development level, family support, medical resources, related behaviors, nursing environment, patients' health behaviors, current medical history, past history, drug use, family history and clinical diagnosis of Alzheimer's patients in inland provinces and cities of China, and made statistics on the related information of patients' health economics. To form a comprehensive assessment of the health economic burden of Alzheimer's disease in China, the primary objectives of the study are as follows:

1. Comprehensively assess the health economic burden of Alzheimer's disease, including medical and non-medical costs.
2. Explore the economic burden of Alzheimer's disease in different stages, including mild cognitive impairment stage, mild to moderate Alzheimer's disease stage and severe Alzheimer's disease stage.
3. To explore the health economic burden of the comorbidity of Alzheimer's disease and other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for selection of centers The study center sample relied on the 192 cognitive centers selected for the 2022 National Health and Health Commission Capacity Building and Continuing Education for Cognitive Impairment Disease Specialty Capacity Building Program.

   The study covered all 31 provincial administrative units in mainland China, divided according to east, center, and west:

   East: Hebei, Beijing, Tianjin, Shandong, Jiangsu, Shanghai, Zhejiang, Fujian, Guangdong, Hainan, Heilongjiang, Jilin, and Liaoning; Central: Henan, Hubei, Hunan, Anhui, Jiangxi, Shanxi; West: Chongqing, Sichuan, Yunnan, Guizhou, Tibet, Shaanxi, Gansu, Qinghai, Xinjiang, Ningxia, Inner Mongolia, Guangxi.
2. amnestic mild cognitive impairment (aMCI) inclusion criteria (all of the following conditions must be met at the same time) and exclusion criteria:

Inclusion criteria:

1. Compliance with Peterson's aMCI diagnostic criteria National Institute on Aging and Alzheimer's Disease Association (NIA-AA) aMCI diagnostic criteria in 2004 [7].
2. Clinical Dementia Rating (CDR) of 0.5.
3. Mini-Mental State Examination (MMSE): ≥17 points on MMSE for those with 0 years of education, ≥20 points for those with less than 7 years, and ≥24 points for those with greater than or equal to 7 years.
4. Memory loss is prominent and may also be accompanied by impairment of other cognitive domains.
5. Insidious onset and slow progression.
6. Not reaching the level of dementia. 3. Alzheimer's disease inclusion criteria (must meet all of the following conditions at the same time) and exclusion criteria:

Inclusion Criteria:

1. Meets the core clinical criteria for probable AD dementia in the 2011 NIA-AA Revised Diagnostic Criteria for AD. [7]
2. Can be categorized as having mild, moderate, or severe Alzheimer's disease.

   1. Mild: progressive cognitive impairment affecting multiple domains and psychobehavioral deficits; significant impact on daily life, primarily impairing instrumental activities, no longer fully independent, occasionally requiring assistance; or a CDR score of 1.0
   2. Moderate: progressive cognitive impairment and psychobehavioral changes; extensive impact on daily life, partial impairment of basic functioning, inability to live independently, frequent need for assistance; or CDR 2.0 score
   3. Severe: progressive cognitive impairment and psychobehavioral changes, may not be able to conduct clinical interviews; severe impact on daily life, impairment of basic activities including self-care, total dependence on help; or CDR 3.0 points
3. CDR greater than 0.5 points.
4. MMSE: <17 points for those with 0 years of education, <20 points for those with less than 7 years, and <24 points for those with greater than or equal to 7 years.
5. Subject has good audiovisual and speech functions or can complete a neuropsychological examination with correction.
6. The subject and the informant can complete relevant examinations and follow-up visits.
7. The subject or his/her authorized delegate signs the informed consent form. 4. Inclusion/exclusion criteria for Alzheimer's disease multiple chronic co-morbidities (aMCI) need to be met in addition to meeting the aMCI inclusion and exclusion criteria or Alzheimer's disease inclusion and exclusion criteria:

Inclusion criteria:

1. Age not less than 60 years
2. Normal or corrected vision and hearing
3. able to provide informed consent signed by him/herself or a legal guardian
4. Newly diagnosed or previously diagnosed with a co-morbid condition other than aMCI or Alzheimer's disease.

Exclusion Criteria:

2. amnestic mild cognitive impairment (aMCI) exclusion criteria: (excluded if any of the following conditions are met):

1. Those with a history of stroke with focal neurologic signs and an imaging presentation consistent with cerebral small vessel disease manifestations (Fazekas score ≥ 2).
2. Presence of mental and neurodevelopmental delays.
3. Presence of other conditions known to cause cognitive impairment.
4. Presence of a disease that prevents cooperation in completing the cognitive examination.
5. Refusal to sign the informed consent form at baseline. 3. Alzheimer's Disease Exclusion Criteria: (Excluded if any of the following criteria are met):

1) Presence of mental and neurodevelopmental delays. 2) Disease that prevents cooperation in completing the cognitive examination. 3) Refusal to sign the informed consent form at baseline. 4. Inclusion/exclusion criteria for Alzheimer's disease multiple chronic co-morbidities (aMCI)

Required on top of meeting aMCI inclusion and exclusion criteria or Alzheimer's disease inclusion and exclusion criteria:

Exclusion Criteria (excluded if any of the following conditions are met):

1. Poor compliance or mental and neurodevelopmental delays.
2. Illness that prevents the completion of the cognitive examination.
3. Refusal to sign an informed consent form at baseline.
4. Severe circulatory, respiratory, urinary, gastrointestinal, hematopoietic diseases (e.g., unstable angina, uncontrolled asthma, active gastric bleeding, etc.) and cancer.
5. No reliably informed person.
6. Patient has a history of alcohol or drug abuse.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research center samples 192 cognitive centers selected by the National Health and Wellness Commission's Capacity Building and Continuing Education for Cognitive Impairment Diseases Project in 2022.
Sampling Method: Non-Probability Sample
Enrollment: 9510 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Direct medical expenses | baseline
  Direct medical expenses refer to the expenses incurred by patients and/or their families for medical and health services related to Alzheimer's disease
Direct non-medical expenses | baseline
  The direct non-medical costs of Alzheimer's disease include care costs, home facilities and repair costs, health care products costs and related expenses incurred during medical treatment. The cost of care includes the salary of caregivers, the expenses of external caregivers, and the travel expenses of caregivers
overhead expenses | baseline
  Indirect costs include the economic loss caused by patients' inability to work, the decrease in the income of informal caregivers, the treatment expenses of caregivers' psychological diseases and the medical expenses incurred by patients with Alzheimer's disease or caregivers due to accidental injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided